CLINICAL TRIAL: NCT06526130
Title: Multiple Sclerosis Comparison of Relapse Incidence After General and Neuraxial Anesthesia: a Retrospective Observational Study
Brief Title: Influence of Anaesthesia Type on Multiple Sclerosis Relapse
Status: Completed | Type: Observational
Sponsor: Varazdin General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 03072024
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; anaesthesia; relapse
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anaesthesia: Intravenous or volatile general anesthesia was preformed with different type of airway management (endotracheal tube, laryngeal mask and bag mask ventilation)
  Interventions: Procedure: General anaesthesia
- Neuraxial anaesthesia: Neuraxial anesthesia was administered using spinal or epidural injections of local anesthetic with or without opioid.
  Interventions: Procedure: Neuraxial anaesthesia

INTERVENTIONS:
Procedure: General anaesthesia — Intravenous or volatile general anesthesia was preformed with different type of airway management (endotracheal tube, laryngeal mask and bag mask ventilation)
  Groups: General anaesthesia
Procedure: Neuraxial anaesthesia — spinal or epidural injections of local anesthetic with or without opioid
  Groups: Neuraxial anaesthesia

SUMMARY:
The influence of anesthesia on the course of multiple sclerosis is poorly investigated and the literature is limited.

The aim of this study is to investigate multiple sclerosis relapse after different types of anesthesia.

DETAILED DESCRIPTION:
The influence of anesthesia on the course of multiple sclerosis is poorly investigated and the literature is limited. A possible relapse after neuraxial anesthesia, it is believed to be associated with local anesthetic's toxicity and concentration.

The aim of this study is to investigate multiple sclerosis relapse after different types of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* multiple sclerosis
* surgical procedure under general anaesthesia
* surgical procedure under neuraxial anaesthesia

Exclusion Criteria:

* patients (medical records) with incomplete data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included adult patientswith multiple sclerosis diagnosis who had undergone general or neuraxial anesthesia in General Hospital Varaždin during the period from 01.01.2012 to 31.12.2022.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Multiple sclerosis relapse after 1 month | 1 month
  Overall incidence of multiple sclerosis relapse after 1 month after anaesthesia
Multiple sclerosis relapse after 3 months | 3 months
  Overall incidence of multiple sclerosis relapse after 3 months after anaesthesia
Multiple sclerosis relapse after 6 months | 6 months
  Overall incidence of multiple sclerosis relapse after 6 months after anaesthesia
Multiple sclerosis relapse after 12 months | 12 months
  Overall incidence of multiple sclerosis relapse after 12 months after anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Monika Kocman Panic, MD, Principal Investigator — Varazdin General Hospital, Varazdin, Croatia

IPD SHARING:
Plan to Share IPD: No